CLINICAL TRIAL: NCT03376919
Title: Efficacy and Usability of the Cyberlegs++ (CLs++) Ortho-prosthesis Modules in Enabling and Enhancing Mobility in Trans-femoral Amputees
Brief Title: The CYBERnetic Lower Limb Cocognitive Ortho-prosthesis Plus Plus, 1st Clinical Study (CLs++)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Fondazione Don Carlo Gnocchi Onlus (Other); Scuola Superiore Sant'Anna di Pisa (Other); Université Catholique de Louvain (Other); University of Ljubljana (Other); Össur Iceland ehf (Industry)
Responsible Party: Principal Investigator, Romain Meeusen, prof, Vrije Universiteit Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VUB-MFYS
Record Dates: First submitted 2017-11-27; First posted 2017-12-19 (Actual); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Lower Limb Amputation Above Knee (Injury)
Keywords: wearable robotics; Unilateral Lower Limb Amputation; gait efficiency
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CLs++ (Experimental): CLs ++ gait training
  Interventions: Device: CLs++ gait training

INTERVENTIONS:
Device: CLs++ gait training — CLs++ gait training

SUMMARY:
The aim of the study is to assess the efficacy and the usability of the cyberlegs ++ ortho prosthesis to improve the mobility and the quality of life in transfemoral amputees . This research focusses on the physical and mental effort needed in locomotion-related tasks and human robot interaction in transfemoral amputees using a novel active prosthesis. This is an international project and foresees 2 clinical studies aimed at assessing the efficacy of the CLs++ modules in different settings.

In this first clinical study, 16 patients with unilateral trans-femoral amputation, 8 at the Vrije Universiteit Brussel Department Human Physiology Research group (VUB-MFYS) and 8 at the Don Gnocchi Foundation, center of Florence.

DETAILED DESCRIPTION:
The aim of the study is to assess the efficacy and the usability of the cyberlegs ++ ortho-prosthesis to improve the mobility and the quality of life in transfemoral amputees. This research focusses on the physical and mental effort needed in locomotion-related tasks and human robot interaction in transfemoral amputees using the CLs++ ortho-prosthesis modules. Unilateral transfemoral amputees will be recruited by a multidisciplinary team (physicians, physiotherapists and psychologists) and a list of inclusion- and exclusions criteria as reported in the 'Eligibility' will be fulfilled to enrol the experiment. If the participant fulfils the requirements to be enrolled, the responsible for the study will provide him/her with the information sheet and will answer all possible questions. Once the participant agrees to participate in the study, he/she will sign the informed consent form and an appointment will also be arranged with the orthopedic workshop to make a spare socket to be used during the clinical testings. In this first clinical study, a set of modules of the three hardware (HW) modules of the CLs++ ortho-prosthesis will be tested, namely the Active Trans-femoral Prosthesis (ATP), the Active Pelvis Orthosis (APO) and the Knee Ankle Foot Orthosis (KAFO).

Each subject will be testing the different combinations of CLs++ modules along with the Wearable Sensory Apparatus (WSA) and the control software (SW):

1)APO+WSA, 2) ATP+WSA, 3) APO+ATP+WSA, 4) APO+KAFO+WSA.

The protocol of the CLs++ first clinical study will be constituted by two main phases:

The initial Phase/familiarization phase:

The appropriate combination of the CL++ modules will be selected based on the clinical evaluation (e.g. walking asymmetry, flexion-extension, hip strenght, strength of the contra-lateral limb) and the subjective feedback in terms of comfort and perceived functionality from the participant. The subjects will be asked to walk at their self-selected speed on a treadmill. To control all variables the functional assessments above will be performed on a treadmill, however, when possible gait related tasks and ancillary tasks will be performed during over-ground walking to asses functional exercise capacity:

* Six Minute Walking Test (6MWT)
* slope walking
* The Timed Up and Go test (TUG) to evaluate balance, Chair standing/sitting.
* The Stair Climbing Test (SCT) to asses stair climbing Electrophysiological and biomechanical parameters will be collected to tell us wether there is an advantage in the use of the novel active prosthetic device in comparison with the current prosthesis only.

The outcomes measures in this study are:

* Electroencephalography (EEG) to record cortical brain activity using an Electro-Encephalography cap (EEGcap, Brain Products GmbH),
* Indirect measurement of the energy expenditure by measuring the oxygen uptake and the produced carbondioxide (ml/min/kg, portable gasanalyzer,Cosmed K5)
* Heart rate (Polar heart rate monitor)

The study foresees the administration of dedicated questionnares to asses the workload such as:

* The Short Form-36 (SF-36) Report of perceived exertion (RPE)-Borg Scale, self-report of the perceived physical effort scale.
* The National Aeronautics and Space Administration task Load indeX (NASA-TLX)
* The System Usability Scale (SUS) to asses the usability of the CLs++ system.
* The SF-36 (short form-36 item) at baseline The subjects will conduct 2 experimental trials during the initial phase, this is with the CLs++ modules and with their current prosthesis only. The participant can rest between the assessments to let the patient recover, with at least 15-30 minutes.

The second phase of the study consist of a intervention, this is a gait training program on the treadmill with the selected combination of CLs++ modules, 1 hour, 3 times a week. Participants will be asked to walk at their self-selected speed and they will be allowed to stop walking whenever they feel tired. At the end of each month we asses wether the experience gained in the training period has effects.

Data of each patient will be analysed separately in order to highlight the occurence of differences between pre- and post- assessment sessions. This is a non-randomized cross-over research, a sample size of 16 subjects will be able to detect a 15% change in walking-related physical effort, in terms of energy expenditure in a single group of trans-femoral amputees with a statistical power >0.9 at the two-sided alpha-level.

ELIGIBILITY:
Inclusion Criteria:

Unilateral trans-femoral amputees both sex age: 30 - 80 yrs Functional K-level 1-4

Exclusion Criteria:

* Severe comorbidity (hemiplegia, degenerative nervous system diseases, severe hip or knee arthrosis,chronic heart failure, chronic obstructive pulmonary, hip or knee replacement, severe sensory deficit
* Pain of the stump/socket poor fitting
* Inability to walk (safely) on a treadmill

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2018-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Energy expenditure | through 6 minutes
  oxygen uptake (ml.kg)/carbondioxide production (ml.kg)

SECONDARY OUTCOMES:
6-Minute Walk Test (6MWT) | through 6 minutes
  the distance (m) walked in 6 minutes, a longer distance represent a better outcome
Timed Up & Go test | through 14 seconds
  the time in seconds the participant needs to stand up out of a chair and walk a 3 meter distance, higher values represent better a better outcome
Sit to stand test | through 5 minutes
  standing up & sitting back down in the chair during 5 minutes, the higher the values the better the results
Slope walking | through 5 minutes
  up and downhill walking
Borg scale-ratings of perceived exertion | minute 6
  subjective measurement, ratings of perceived exertion, numeric scale that ranges between 6 (no exertion at all) and 20 (maximal exertion). 7= extremely light, 9 = very light, 11=light, 13=somewhat hard, 15=hard, 17=very hard, 19=Extremely hard. A higher score is a worse outcome
National Aeronautics & Space Administration Task Load Index | minute 6
  Subjective rating scale
Short Form 36 questionnaire | minute 1
  subjective measurement
Prosthesis Evaluation Questionnaire | up to 24 weeks
  subjective evaluation of the prosthesis
System Usability Scale | up to 24 weeks
  subjective evaluation of the new prosthesis
Stair Climbing test | through 5 minutes
  the possibility to ascent and descent stairs
EEG | through 6 minutes
  electro-encephalography

IPD SHARING:
Plan to Share IPD: No